CLINICAL TRIAL: NCT00429806
Title: DHEA Bioavailability Following Administration of Vaginal Suppositories in Post-Menopausal Women With Vaginal Atrophy-Phase I Randomized,Placebo-Controlled, Double-Blind Study.
Brief Title: DHEA Bioavailability Following Administration of Vaginal Suppositories in Post-Menopausal Women With Vaginal Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-213
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Vaginal Atrophy
Keywords: Vaginal atrophy; DHEA; Prasterone; Menopause
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo suppository; once daily for 7 days.
  Interventions: Drug: Placebo
- DHEA 0.50% (Experimental): DHEA 0.50% (6.5 mg) suppository; once daily for 7 days.
  Interventions: Drug: DHEA
- DHEA 1.0% (Experimental): DHEA 1.0% (13 mg) suppository; once daily for 7 days.
  Interventions: Drug: DHEA
- DHEA 1.8% (Experimental): DHEA 1.8% (23.4 mg) suppository; once daily for 7 days.
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: DHEA — DHEA
  Other Names: dehydroepiandrosterone; prasterone
  Arms: DHEA 0.50%; DHEA 1.0%; DHEA 1.8%
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the systemic bioavailability of DHEA and its metabolites and the pharmacokinetics of vaginal suppositories at four different DHEA concentration.

DETAILED DESCRIPTION:
Humans, are unique among animal species in having adrenals that secrete large amounts of the inactive precursor steroids dehydroepiandrosterone (DHEA) and especially its sulfate DHEA-S. The marked reduction in the formation of DHEA-S by the adrenals during aging results in a dramatic fall in the formation of androgens and estrogens in peripheral target tissues, a situation that has been proposed to be associated with age-related diseases including skin atrophy, insulin resistance and obesity. Much attention has been given to the benefits of DHEA administered to postmenopausal women, especially on the bone, skin, vagina and well being after oral as well as percutaneous administration of the precursor steroid.

Therefore, this study proposes to evaluate the systemic bioavailability and the effectiveness of 1.3 mL vaginal suppositories of DHEA at 4 different concentrations (0.0%, 0.5%, 1.0% et 1.8%) following 1 week administration of vaginal suppositories in post-menopausal women with vaginal atrophy. This is a phase I, randomized, placebo-controlled, double-blind study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women,
* Experiencing one symptom of vaginal atrophy (vaginal dryness, vaginal and/or vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity or vaginal bleeding associated with sexual activity,
* Women having a low maturation index and a vaginal pH above 5,
* Endometrial thickness of 4 mm or less at transvaginal ultrasonography,
* Body weight within 18.5 and 32.0 according to body mass index.

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding,
* Active or history of thromboembolic disease,
* Significant metabolic or endocrine disease,
* Significant complication on previous hormonal therapy,
* Use of hormonal implants within 6 months prior to study entry,
* Use of oral estrogen, progestin or DHEA in the 8 weeks prior to baseline,
* Use of natural (phytoestrogens) or herbal products in the 2 weeks prior to baseline,
* Chronic use of corticosteroids,
* Hypertension not controlled by standard therapy.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The evaluation of the systemic bioavailability of DHEA and its metabolites. | Day 1-2 and Day 7-8
The pharmacokinetics of vaginal suppositories at four different DHEA concentrations. | Day 1-2 and Day 7-8

SECONDARY OUTCOMES:
The safety and tolerance of the suppositories. | Day 1 to Day 8 (plus follow-up of Adverse Events for 30 days after last dose)
The effect of treatment on maturation index and value | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Fernand Labrie, MD, Ph D, Study Chair — CHUL Research Center Director; Cusan Leonello, MD Ph D, Principal Investigator — CHUL Research Center
Locations (1):
- Clinique des traitements hormonaux CHUL Research Center, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Labrie F, Cusan L, Gomez JL, Cote I, Berube R, Belanger P, Martel C, Labrie C. Effect of intravaginal DHEA on serum DHEA and eleven of its metabolites in postmenopausal women. J Steroid Biochem Mol Biol. 2008 Sep;111(3-5):178-94. doi: 10.1016/j.jsbmb.2008.06.003. Epub 2008 Jun 12. PMID 18598765
- [Result] Labrie F, Martel C, Berube R, Cote I, Labrie C, Cusan L, Gomez JL. Intravaginal prasterone (DHEA) provides local action without clinically significant changes in serum concentrations of estrogens or androgens. J Steroid Biochem Mol Biol. 2013 Nov;138:359-67. doi: 10.1016/j.jsbmb.2013.08.002. Epub 2013 Aug 14. PMID 23954500
- [Result] Labrie F, Martel C. A low dose (6.5 mg) of intravaginal DHEA permits a strictly local action while maintaining all serum estrogens or androgens as well as their metabolites within normal values. Horm Mol Biol Clin Investig. 2017 Feb 1;29(2):39-60. doi: 10.1515/hmbci-2016-0042. PMID 27997350